CLINICAL TRIAL: NCT02439281
Title: ROPIVACAINE WITH CLONIDINE FOR PEDIATRIC RECTUS SHEATH BLOCKS- THE MAGIC COMBINATION? - A Double Blinded Prospective Study
Brief Title: Ropivacaine With Clonidine For Pediatric Rectus Sheath Blocks- The Magic Combination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patients were discharged on the day of the surgery.
Sponsor: Mihaela Visoiu (Other)
Responsible Party: Sponsor-Investigator, Mihaela Visoiu, Director Acute Interventional Perioperative Pediatric Pain Service, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO14100075
Record Dates: First submitted 2015-04-16; First posted 2015-05-08 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
Keywords: Ropivacaine; Anesthesia adjuncts; clonidine; laparoscopic appendectomy; rectus sheath block
MeSH Terms: conditions — Pain, Postoperative | interventions — Clonidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine Group (Active Comparator): Ropivacaine Group will receive ropivacaine 0.5% (10 ml) injected bilaterally in the posterior rectus sheath, at the umbilicus location.
  Interventions: Drug: Ropivacaine
- Ropivacaine/ Clonidine Group (Experimental): Ropivacaine/ Clonidine Group will receive ropivacaine 0.5% (10 ml) and clonidine (2mcg/kg) injected bilaterally in the posterior rectus sheath, at the umbilicus location.
  Interventions: Drug: Clonidine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Clonidine — Only the Ropivacaine /clonidine group will receive clonidine (2mcg/kg) injected with ropivacaine.
  Other Names: kapvay; Catapres; Duraclon; Nexiclon
  Arms: Ropivacaine/ Clonidine Group
Drug: Ropivacaine — One hundred pediatric patients (10-17 years old) scheduled for laparoscopic appendectomy will be randomized to the two treatment groups: the Ropivacaine Group will receive ropivacaine 0.5% (10 ml) injected bilateral in Both groups will receive ropivacaine 0.5% (10 ml) injected bilaterally for the rectus sheath block
  Other Names: Naropin

SUMMARY:
Background: Millions of pediatric patients undergo laparoscopic surgeries every year and many of them suffer significant pain and anxiety. Patient's anxiety correlates with the severity of pain and effective postoperative analgesia is necessary for optimal recovery. Single injections ultrasound guided rectus sheath blocks provide satisfactory postoperative analgesia after pediatric laparoscopic appendectomy, however they are short lived. Searching for a blocking agent that last long enough to outlast pain and has minimal side effects is a difficult task. Using a combination of drugs yielded mixed results. Few pediatric studies showed at best a weak trend in favor of clonidine prolonging analgesia after some blocks, but anxiolytic properties of clonidine were not investigated. This study will compare rectus sheath ropivacaine blocks with ropivacaine and clonidine blocks.

Methods: One hundred pediatric patients (10-17 years old) scheduled for laparoscopic appendectomy will be double blinded and randomized to the two treatment groups: the Ropivacaine Group will receive ropivacaine 0.5% (10 ml) injected bilaterally in the posterior rectus sheath, at the umbilicus location, and Ropivacaine Clonidine Group will receive ropivacaine 0.5% (10 ml) and clonidine (2mcg/kg). Post-operative analgesia will be provided with ketorolac and acetaminophen around the clock, and morphine, or/and oxycodone as needed. The primary aim is to determine if ropivacaine combined with clonidine prolongs duration of paresthesia. The secondary aims are to determine if the use of clonidine decreases anxiety level, prolongs duration of analgesia, and decreases pain severity at umbilicus laparoscopic site, reduces the need for analgesics, improves satisfaction with pain control, and is associated with complications such as oversedation, hypotension, and bradycardia.

Conclusions: Every hour of excellent analgesia count and a prolongation of block duration by at least 50% is clinical relevant. The investigators hypothesize that rectus sheath injections with ropivacaine and clonidine offer improved pain management compared to ropivacaine alone.

DETAILED DESCRIPTION:
Objective: The primary aim is to determine if ropivacaine combined with clonidine prolongs duration of paresthesia at the umbilicus. The secondary aims are to determine if the use of clonidine decreases anxiety level, prolongs duration of analgesia, decreases pain severity at the umbilicus laparoscopic site, reduces the need for pain medication, improves satisfaction with pain control, and is associated with complications such as oversedation, hypotension, and bradycardia.

Specific Aims: Aim 1 will determine if the duration of sensory block (paresthesia) after ultrasound guided single injections rectus sheath blocks performed with ropivacaine/ clonidine is longer than duration of paresthesia after rectus sheath blocks performed with ropivacaine alone. The investigators hypothesize that rectus sheath injections with ropivacaine and clonidine result in longer duration of sensory block (paresthesia) compared to ropivacaine alone.

Aim 2 will determine if the use of clonidine decreases postoperative anxiety scores and if postoperative pain scores correlate with anxiety scores. The investigators hypothesize that patient postoperative anxiety scores are lower in the Ropivacaine/Clonidine group and postoperative anxiety scores decrease more in Ropivacaine /Clonidine Group, than in the Ropivacaine Group. The investigators expect that preoperative and postoperative Numeric Rating Scale(NRS) scores reported by the patient will correlate moderately (0.3-0.49) to high (equal /or >0.5) with preoperative and postoperative anxiety level.

Aim 3 will determine if rectus sheath injections with ropivacaine/ clonidine prolongs duration of analgesia at umbilicus instrument site, decreases analgesic consumption, improves satisfaction with pain control, and has minimal complications such as oversedation, bradycardia, and hypotension. The investigators hypothesize that rectus sheath injections with ropivacaine/ clonidine would result in longer duration of analgesia compared to ropivacaine alone, lower pain scores at umbilicus, less need for pain medication consumption for pain at umbilicus and for the first 18 hours, better satisfaction with pain control from patient, parent and nurse. The investigators expect no difference in incidence of oversedation, hypotension, and bradycardia episodes.

Background: Millions of pediatric patients undergo laparoscopic surgeries every year and many of them suffer significant pain on the day of surgery and the subsequent days. Pain is a sensory and emotional experience, modified by multiple factors, including anxiety. Patient's anxiety correlates with the severity of pain. Children that are very anxious before surgery have been found to have more postoperative pain, delayed hospital discharge, higher incidence of emergence delirium, sleep disturbances, and other maladaptive behavior changes that can last up to a few weeks following surgery. Laparoscopic appendectomy can cause significant pain and anxiety despite the minimally invasive approach. The investigators' recent completed prospective study showed that on the day after surgery, pain after laparoscopic appendectomy correlated very well with postoperative anxiety scores (Pearson coefficient =0.539; pending publication results from 133 subjects, 11-17 years old, that underwent laparoscopic appendectomy).

Effective postoperative analgesia after laparoscopic appendectomy is necessary for optimal recovery. A multimodal approach includes regional analgesia techniques, improves analgesia, and reduces side-effects from opioids use. Unfortunately, pain associated with this procedure extends after the day of surgery. Continuous peripheral nerve blocks can be effective, but are deemed excessively invasive in the context of this minimally invasive surgery. Single injection nerve blocks are appropriate, but the duration with a long acting local anesthetic is only around 12 hours, and do not match the most painful part of postoperative period, the first 24 hours. Over the last years, the challenge of developing a blocking agent that lasts long enough to outlast pain and has minimal side effects has been addressed by combining different drugs (epinephrine, clonidine, dexamethasone, tramadol, buprenorphine, midazolam, magnesium, dexmedetomidine, and ketamine) and yielded mixed results. Among these, clonidine, an alpha 2 adrenoreceptor agonist has been shown to prolong the duration of analgesia when administered in epidural space in children. Clonidine has also been added to local anesthetic for peripheral nerve blocks but its perineural use is controversial and the exact mechanism is unclear. Its action is not entirely attributed to an alpha -adrenergic effect at the nerve; rather, it is possibly secondary to the blockade of the current through hyperpolarization- activated cyclic nucleotide-gated channels, resulting in the enhancement of activity-dependent hyperpolarization.

From the limited available data, perineurally administered clonidine appears to be safe, but the results remain controversial. Adult metaanalysis have found that clonidine from 30-300 mcg prolongs the time to the first analgesic request by only 2-2.5 hrs. Furthermore, clonidine prolonged sensory and motor blockade with all local anesthetic except mepivacaine.

The pediatric literature regarding the use of clonidine for peripheral nerve blocks lags behind adult literature and is conflicting. Few small and under-powered studies showed at best a weak trend in favor of clonidine. A retrospective review of 215 patients showed that the use of clonidine prolongs the duration of infraclavicular, lumbar plexus, femoral, fascia iliaca and sciatic nerve blocks by 20-50%. However, the prolongation is block location dependent, and increased the incidence of motor block. This effect was only seen with diluted concentrations of bupivacaine 0.125% and ropivacaine 0.2%. No pediatric or adult studies were performed involving trunk blocks such as rectus sheath, transversus abdominis plane, or paravertebral nerve blocks.

Side effects reported after clonidine was administered neuraxially or perineurally are hypotension, sedation, fainting, and prolonged motor blockade. Hypotension and sedation appear to be limited up to doses of 150 mcg. However, Petroheilou et al. reported intraoperatively hemodynamic stability after administration of clonidine at 3 mcg/kg. Clonidine 1-2 mcg/kg is suggested for use with local anesthetic for single injections peripheral nerve blocks.

Clonidine can help to relieve postoperative anxiety, and subsequently improve pain control. Minimal sedation after clonidine administration can be desired for some pediatric patients. Clonidine at 2 mcg/kg prevents sevoflurane-induced agitation and can be used as premedication in children. No studies have investigated its role as an anxiolytic when added to local anesthetic for a nerve block.

The Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center (CHP of UPMC) has a dedicated service to provide regional anesthesia techniques and performs peripheral nerve blocks on a regular basis. Over the last academic year, 190 patients that underwent laparoscopic appendectomy had peripheral nerve blocks (rectus sheath and transversus abdominis plane) performed for pain control. Children localized the majority of their pain to the umbilicus instrument site. This pain interferes with patients' activities such as ambulation, eating, and bedside activities. The principal investigator performed a retrospective chart review to compare postoperative analgesia from rectus sheath blocks and a combination of transversus abdominis plane and rectus sheath blocks. The postoperative opioid consumption and pain scores were similar. Since then, the primary investigator performs only ultrasound guided rectus sheath blocks for postoperative analgesia after laparoscopic appendectomy. A recent pediatric study showed that the rectus sheath blocks in combination with multimodal analgesia are effective for postoperative pain control after mentioned procedure. Unfortunately the duration of these blocks performed with maximum 20 ml of bupivacaine 0.25% with adrenaline did not outlast the most painful period. The investigators believe that rectus sheath blocks with ropivacaine 0.5% and clonidine (2 mcg/kg) will prolong the duration of blocks, can reduce postoperative pain and anxiety, facilitate discharge, and decrease unplanned hospital admission secondary to pain, and can contribute to an increased patient and family satisfaction, and decrease costs for the hospital, insurer, and the patient.

Significance: To the investigators' knowledge, this is the first study to investigate whether ropivacaine /clonidine rectus sheath blockade is a better and more complete therapeutic regimen for patients undergoing laparoscopic appendectomy. While the patients that underwent uncomplicated laparoscopic appendectomy are treated as inpatient for at least one day, CHP wants to implement early discharge strategies. Unfortunately, the pain after day of surgery can be significant and some parents can be reluctant to have their children discharged. The analgesia advices can be poorly retained. The parents can feel overwhelmed about home pain management. Some parents believe that using pain medication in childhood may lead to later drug abuse. This is concerning as parents often undermedicate their child's pain, with up to 60% of parents administering less than the prescribed analgesia on the following day after surgery discharge. A child with long lasting pain control and less anxiety from ropivacaine/clonidine rectus sheath blockade will help the parent cope with the surgical event, and can facilitate early discharge.

Additionally, patient's satisfaction with pain control is becoming an increasingly important aspect of health care reimbursements reported via the Hospital Assessment of Healthcare Providers and Systems (HCAHPS) survey. The ropivacaine/ clonidine rectus sheath blockade in combination with multimodal therapy can be better therapeutic regimen that standard of care, and can improve quality of care, increase satisfaction and save health care costs.

ELIGIBILITY:
Inclusion Criteria:

* age 10-17 years
* scheduled for elective laparoscopic appendectomy
* weight >/=34kg
* complete postoperative questionnaires.

Exclusion Criteria:

* patients younger than 10 years and 18 years or older
* weight < 34 kg
* weight >/=100 kg
* patient and family refusal
* non-English-speaking patients and families
* cognitive impairment
* developmental delay
* allergies to medications used in the study (hydromorphone, oxycodone, acetaminophen, ketorolac, ropivacaine, and clonidine)
* need for opioids via patient controlled analgesia device
* patients with a positive pregnancy test
* local infection at planned injection sites
* patients with failed rectus sheath blocks
* patients that require opioids via patient controlled analgesia device
* patients with laparoscopic procedure converted to open
* patients that will not be able to place the time of return to normal sensation within 1 hour of its occurrence
* patients with no follow up possible
* the patients that will be discharged home before the resolution on paresthesia will be excluded from analysis of the first aim.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Visoiu, MD, Principal Investigator — Children's Hospital of UPMC
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groenewald CB, Rabbitts JA, Schroeder DR, Harrison TE. Prevalence of moderate-severe pain in hospitalized children. Paediatr Anaesth. 2012 Jul;22(7):661-8. doi: 10.1111/j.1460-9592.2012.03807.x. Epub 2012 Feb 15. PMID 22332912
- [Background] Hegarty M, Calder A, Davies K, Shave M, Christiansen E, Meyer T, von Ungern-Sternberg BS. Does take-home analgesia improve postoperative pain after elective day case surgery? A comparison of hospital vs parent-supplied analgesia. Paediatr Anaesth. 2013 May;23(5):385-9. doi: 10.1111/pan.12077. Epub 2012 Nov 20. PMID 23167309
- [Background] Tsao JC, Lu Q, Myers CD, Kim SC, Turk N, Zeltzer LK. Parent and child anxiety sensitivity: relationship to children's experimental pain responsivity. J Pain. 2006 May;7(5):319-26. doi: 10.1016/j.jpain.2005.12.004. PMID 16632321
- [Background] Tsao JC, Meldrum M, Kim SC, Zeltzer LK. Anxiety sensitivity and health-related quality of life in children with chronic pain. J Pain. 2007 Oct;8(10):814-23. doi: 10.1016/j.jpain.2007.05.011. Epub 2007 Jul 5. PMID 17613277
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Liu Y, Seipel C, Lopez ME, Nuchtern JG, Brandt ML, Fallon SC, Manyang PA, Tjia IM, Baijal RG, Watcha MF. A retrospective study of multimodal analgesic treatment after laparoscopic appendectomy in children. Paediatr Anaesth. 2013 Dec;23(12):1187-92. doi: 10.1111/pan.12271. Epub 2013 Sep 25. PMID 24112856
- [Background] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Background] Bailard NS, Ortiz J, Flores RA. Additives to local anesthetics for peripheral nerve blocks: Evidence, limitations, and recommendations. Am J Health Syst Pharm. 2014 Mar 1;71(5):373-85. doi: 10.2146/ajhp130336. PMID 24534592
- [Background] Akin A, Ocalan S, Esmaoglu A, Boyaci A. The effects of caudal or intravenous clonidine on postoperative analgesia produced by caudal levobupivacaine in children. Paediatr Anaesth. 2010 Apr;20(4):350-5. doi: 10.1111/j.1460-9592.2010.03259.x. Epub 2010 Feb 11. PMID 20158620
- [Background] Rochette A, Troncin R, Raux O, Dadure C, Lubrano JF, Barbotte E, Capdevila X. Clonidine added to bupivacaine in neonatal spinal anesthesia: a prospective comparison in 124 preterm and term infants. Paediatr Anaesth. 2005 Dec;15(12):1072-7. doi: 10.1111/j.1460-9592.2005.01664.x. PMID 16324026
- [Background] Kroin JS, Buvanendran A, Beck DR, Topic JE, Watts DE, Tuman KJ. Clonidine prolongation of lidocaine analgesia after sciatic nerve block in rats Is mediated via the hyperpolarization-activated cation current, not by alpha-adrenoreceptors. Anesthesiology. 2004 Aug;101(2):488-94. doi: 10.1097/00000542-200408000-00031. PMID 15277933
- [Background] McCartney CJ, Duggan E, Apatu E. Should we add clonidine to local anesthetic for peripheral nerve blockade? A qualitative systematic review of the literature. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):330-8. doi: 10.1016/j.rapm.2007.02.010. PMID 17720118
- [Background] Popping DM, Elia N, Marret E, Wenk M, Tramer MR. Clonidine as an adjuvant to local anesthetics for peripheral nerve and plexus blocks: a meta-analysis of randomized trials. Anesthesiology. 2009 Aug;111(2):406-15. doi: 10.1097/ALN.0b013e3181aae897. PMID 19602964
- [Background] Petroheilou K, Livanios S, Zavras N, Hager J, Fassoulaki A. Sciatic lateral popliteal block with clonidine alone or clonidine plus 0.2% ropivacaine: effect on the intra-and postoperative analgesia for lower extremity surgery in children: a randomized prospective controlled study. BMC Anesthesiol. 2012 Feb 1;12:2. doi: 10.1186/1471-2253-12-2. PMID 22297020
- [Background] Trifa M, Ben Khalifa S, Jendoubi A, Zribi N, Regaya T, Engelhardt T. Clonidine does not improve quality of ropivacaine axillary brachial plexus block in children. Paediatr Anaesth. 2012 May;22(5):425-9. doi: 10.1111/j.1460-9592.2012.03809.x. Epub 2012 Feb 6. PMID 22309507
- [Background] Dagher C, Yazigi A, Rkaibe N. Clonidine as adjuvant for bupivacaine in ilioinguinal block does not prolong postoperative analgesia in pediatric and also in adult patients. Paediatr Anaesth. 2006 Feb;16(2):224-5; author eply 225. doi: 10.1111/j.1460-9592.2005.01809.x. No abstract available. PMID 16430430
- [Background] Cucchiaro G, Ganesh A. The effects of clonidine on postoperative analgesia after peripheral nerve blockade in children. Anesth Analg. 2007 Mar;104(3):532-7. doi: 10.1213/01.ane.0000253548.97479.b8. PMID 17312203
- [Background] Ivani G, Conio A, De Negri P, Eksborg S, Lonnqvist PA. Spinal versus peripheral effects of adjunct clonidine: comparison of the analgesic effect of a ropivacaine-clonidine mixture when administered as a caudal or ilioinguinal-iliohypogastric nerve blockade for inguinal surgery in children. Paediatr Anaesth. 2002 Oct;12(8):680-4. doi: 10.1046/j.1460-9592.2002.00935.x. PMID 12472703
- [Background] Kaabachi O, Zerelli Z, Methamem M, Abdelaziz AB, Moncer K, Toumi M. Clonidine administered as adjuvant for bupivacaine in ilioinguinal-iliohypogastric nerve block does not prolong postoperative analgesia. Paediatr Anaesth. 2005 Jul;15(7):586-90. doi: 10.1111/j.1460-9592.2005.01497.x. PMID 15960643
- [Background] Sharpe P, Klein JR, Thompson JP, Rushman SC, Sherwin J, Wandless JG, Fell D. Analgesia for circumcision in a paediatric population: comparison of caudal bupivacaine alone with bupivacaine plus two doses of clonidine. Paediatr Anaesth. 2001 Nov;11(6):695-700. doi: 10.1046/j.1460-9592.2001.00748.x. PMID 11696146
- [Background] Lonnqvist PA. Adjuncts should always be used in pediatric regional anesthesia. Paediatr Anaesth. 2015 Jan;25(1):100-6. doi: 10.1111/pan.12526. Epub 2014 Sep 17. PMID 25230242
- [Background] Kulka PJ, Bressem M, Tryba M. Clonidine prevents sevoflurane-induced agitation in children. Anesth Analg. 2001 Aug;93(2):335-8, 2nd contents page. PMID 11473855
- [Background] Mukherjee A, Das A, Basunia SR, Chattopadhyay S, Kundu R, Bhattacharyya R. Emergence agitation prevention in paediatric ambulatory surgery: A comparison between intranasal Dexmedetomidine and Clonidine. J Res Pharm Pract. 2015 Jan-Mar;4(1):24-30. doi: 10.4103/2279-042X.150051. PMID 25710047
- [Background] Nishina K, Mikawa K. Clonidine in paediatric anaesthesia. Curr Opin Anaesthesiol. 2002 Jun;15(3):309-16. doi: 10.1097/00001503-200206000-00006. PMID 17019218
- [Background] Bergendahl H, Lonnqvist PA, Eksborg S. Clonidine in paediatric anaesthesia: review of the literature and comparison with benzodiazepines for premedication. Acta Anaesthesiol Scand. 2006 Feb;50(2):135-43. doi: 10.1111/j.1399-6576.2006.00940.x. PMID 16430532
- [Background] Hamill JK, Liley A, Hill AG. Rectus sheath block for laparoscopic appendicectomy: a randomized clinical trial. ANZ J Surg. 2015 Dec;85(12):951-6. doi: 10.1111/ans.12950. Epub 2015 Jan 12. PMID 25581711
- [Background] Spielberger Charles Donald ECD. State-trait Anxiety Inventory for Children: STAIC : How I Feel Questionnaire : Professional Manual 1973.
- [Background] Fortier MA, Kain ZN. Treating perioperative anxiety and pain in children: a tailored and innovative approach. Paediatr Anaesth. 2015 Jan;25(1):27-35. doi: 10.1111/pan.12546. Epub 2014 Sep 30. PMID 25266082
- [Background] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Background] Hamers JP, Abu-Saad HH. Children's pain at home following (adeno) tonsillectomy. Eur J Pain. 2002;6(3):213-9. doi: 10.1053/eujp.2001.0326. PMID 12036308
- [Derived] Visoiu M, Scholz S, Malek MM, Carullo PC. The addition of clonidine to ropivacaine in rectus sheath nerve blocks for pediatric patients undergoing laparoscopic appendectomy: A double blinded randomized prospective study. J Clin Anesth. 2021 Aug;71:110254. doi: 10.1016/j.jclinane.2021.110254. Epub 2021 Mar 19. PMID 33752119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Group | Ropivacaine/ Clonidine Group
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 patient withdrew the consent and one surgery was cancelled but these 2 patients were included in age , gender , weight and demographics. Blocks done on only 48 Only the patients that had the time when the numbness went away were compared
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Group | Ropivacaine/ Clonidine Group | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 26 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 13. [11.50 to 15.50] | 13 [11 to 15] | 13 [11 to 15.50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
preoperative anxiety [Median (Inter-Quartile Range); unit: units on a scale] — To measure anxiety , the participants completed the state version of the State-Trait Anxiety Inventory for Children . This scale consists of 20 statements that ask the patient how they feel at that particular moment (e.g., "I feel…"), by checking one of the three alternatives that describe the child best (e.g., "very calm," "calm," or "not calm"). The total score for this scale ranges from 20-60. The highest number means more anxiety, worse outcome Only patients with completed scale were included Population: data was available only for the patients listed, 21, respectively 24 in each group
  units on a scale
    number analyzed (Participants) | 21 | 24 | 45
    (all) | 33 [31 to 39] | 39 [31.5 to 45] | 35 [31 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Block (Paresthesia)
Description: The investigators hypothesize that rectus sheath injections with ropivacaine and clonidine result in longer duration of sensory block (paresthesia) compared to ropivacaine alone.
Time Frame: Indicated by return of normal sensation (expected average of 12 hours after block placement).
Population: only patients that were able to report the time when the numbness went away were analysed and compared
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
Number analyzed (Participants) | 20 | 17
minutes | 823.5 [509.50 to 1080] | 540 [360 to 1015]
Statistical Analysis 1: Comparison: Ropivacaine/ Clonidine Group vs Ropivacaine Group; Test type: Other; p = 0.4510, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Satisfaction With Pain Control From Patient
Description: The investigators hypothesize that rectus sheath injections with ropivacaine/ clonidine would result in better satisfaction with pain control.
Time Frame: Prior to hospital discharge (up to 24 hours after surgery)
Population: only patients with satisfaction scores documented and other inclusion criteria met were analysed and compared; A numeric satisfaction scale 1-10 ( 1 not satisfied, 10 being very satisfied) was used
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
Number analyzed (Participants) | 20 | 16
units on a scale | 9 [9 to 10] | 9 [8 to 10]
Statistical Analysis 1: Comparison: Ropivacaine/ Clonidine Group vs Ropivacaine Group; Test type: Other; p = 0.8914, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Complications Rate
Description: The investigators expect no difference in incidence of complications (e.g. oversedation, hypotension, bradycardia episodes, etc.).
Time Frame: until study completion
Population: The patients that received a nerve block were analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
Number analyzed (Participants) | 25 | 24
Participants | 1 | 1

4. Secondary Outcome: Change in Anxiety Scores
Description: The investigators hypothesize that patient postoperative anxiety scores are lower in the Ropivacaine/Clonidine group and postoperative anxiety scores decrease more in Ropivacaine /Clonidine Group, than in Ropivacaine Group.
Time Frame: 6 hours after block placement
Population: Only patients that a completed anxiety scale were analyzed . State-Trait Anxiety Inventory for Children consists of 20 statements; how they feel at that particular moment ( "I feel…"), by checking one of the three alternatives that describe the child best "very calm," "calm," or "not calm"). The total score ranges from 20-60 ( worse outcome).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine Group | Ropivacaine/ Clonidine Group
Number analyzed (Participants) | 18 | 23
units on a scale | 30 [27 to 30] | 29 [26 to 32]

5. Secondary Outcome: Duration of Analgesia at Umbilicus Instrument Site-How Many Minutes Passed From the Time When the Blocks Where Performed Until Patient Reported Pain at Umbilicus
Description: The investigators hypothesize that rectus sheath injections with ropivacaine/ clonidine would result in longer duration of analgesia and decreased pain scores compared to ropivacaine alone.
Time Frame: indicated by the first request for pain medication at umbilicus site
Population: only patients with documented duration of numbness and documented first pain scores at umbilicus were included in analysis of this secondary outcome
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
Number analyzed (Participants) | 16 | 15
minutes | 230 [137.50 to 388.00] | 240 [144 to 359]
Statistical Analysis 1: Comparison: Ropivacaine/ Clonidine Group vs Ropivacaine Group; Test type: Other; p = 0.9531, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Average Pain Severity at the Umbilicus Laparoscopic Site
Description: Numeric Rating Pain Scores ( 0-10), will be obtained every 2 hours after PACU discharge up to 18 hours or until hospital discharge, whichever occurs first. The pain score of 0, means no pain, is a good outcome , and a pain score of 10 is excruciating pain, a very bad outcome. The average of these scores will be evaluated.The pain scores will not longer be documented after the numbness went away.
Time Frame: Logistic regression of the 4 th pain score assessment
Population: Only patients with available average pain scores at the 4 th pain assessment were compared.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine Group | Ropivacaine/ Clonidine Group
Number analyzed (Participants) | 19 | 18
units on a scale | 2 [0 to 2] | 1.5 [0 to 4]
Statistical Analysis 1: Comparison: Ropivacaine Group vs Ropivacaine/ Clonidine Group; Test type: Other; p = 0.7780, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Medication Consumption
Description: Total intravenous morphine equivalents mg/kg
Time Frame: 18 hours after surgery
Population: Only patients with successful blocks were included. Two patients were deemed to have incomplete/ failed blocks and 2 patients did not have any blocks.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
Number analyzed (Participants) | 25 | 21
mg/kg | 0.20 [0.17 to 0.24] | 0.22 [0.15 to 0.36]
Statistical Analysis 1: Comparison: Ropivacaine/ Clonidine Group vs Ropivacaine Group; Test type: Other; p = 0.5692, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: through study completion, an average 36 hours
Description: Only patients that underwent the rectus sheath blocks were included in the adverse report description. Two patients were included in the study, but after randomization, 1 surgery was canceled, and another one was withdrew by the father. These 2 patients did not underwent any blocks
Arm/Group | Ropivacaine/ Clonidine Group | Ropivacaine Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

LIMITATIONS AND CAVEATS:
I had to stop the study after 50 patients because the patients that underwent laparoscopic appendectomy were sent home on a day of surgery, before the numbness wore off.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02439281/Prot_SAP_000.pdf